CLINICAL TRIAL: NCT03983421
Title: Feasibility of an Early Detection Program for Early Psychosis on a College Campus
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-174; 1R34MH120777-01 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-06-12 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Psychosis; First Episode Psychosis; Clinical High Risk for Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students Enrolled In Coordinated Specialty Care: The number of students determined eligible for Coordinated Specialty Care that were originally screened through the PQ-B at the college counseling center.

SUMMARY:
The objective of the proposed study is to determine the feasibility of an Early Detection program that aims to: (i) identify college students at clinical high risk (CHR) of psychosis or with first episode psychosis (FEP), and (ii) efficiently link them to coordinated specialty care (CSC) services for a 2nd stage screen, a clinical assessment, and appropriate treatment. The study will also determine pathways to care and perceived barriers to care among those students enrolled in Coordinated Specialty Care.

DETAILED DESCRIPTION:
Long duration of untreated psychosis (DUP) is associated with poor outcomes, including higher rates of suicide, hospitalization, and overall low functioning. More widespread use of effective strategies to decrease DUP are needed to address the substantial discrepancy between the actual (i.e., on average 2 years) and recommended time (i.e., 3 months) between the appearance of psychotic symptoms and the initiation of treatment. Early detection (ED) programs aim to decrease DUP by increasing case identification and removal of barriers to coordinated specialty care (CSC). The most studied components of ED programs include: (i) educational campaigns; ED response teams designed to optimize the referral processes to CSC; and to a lesser extent, screening among high-risk groups. While results of studies on individual ED components have been inconsistent, combinations of ED components have had more success in reducing DUP. For example, the Treatment and Intervention in Psychosis ED program, which included educational campaigns and ED teams, reported an average decrease in DUP from 1.5 years to 0.5 years pre-post implementation. The evidence on community-based ED programs is large and growing but very little is known about the effectiveness of ED services on college campuses in the United States. This gap in the literature is problematic because, with the first symptoms of psychosis being most likely to surface among college age young adults, college campuses are critical locations to identify and refer individuals to CSC who are at increased risk of first episode psychosis (FEP). The investigators aim to address this gap in the literature.

The long-term goal of this program of research is to improve clinical and functional outcomes among college students with early stages of psychosis by reducing DUP. The objective of the proposed study is to determine the feasibility of an ED program that aims to: (i) identify college students at CHR of psychosis or with FEP, and (ii) efficiently link them to CSC services for a 2nd stage screen and a clinical assessment among those determined eligible. Students will be referred to treatment based on the results of the assessment (the University of New Mexico Department of Psychiatry CSC program includes clinical services for both FEP and CHR).

The study will also determine pathways to care and perceived barriers to care among those students enrolled in Coordinated Specialty Care.

ELIGIBILITY:
Inclusion Criteria:

1. 15-30 year-old college students who present to the University of New Mexico (UNM) Early Program or the UNM CONNECT program for an intake,
2. screen positive for clinical high risk on the Structured Interview for Prodromal Syndromes (SIPS) or first episode psychosis on the Structured Clinical Interview for Diagnostic Statistical Manual IV
3. agree to participate in the study.

Exclusion Criteria:

1. below the age of 15 years old or above the age of 30,
2. not UNM college students,
3. screen negative for clinical high risk or first episode psychosis,
4. refuse to participate in the study,
5. cognitively unable to provide informed consent as demonstrated by a brief cognitive screen prior to completion of the enrollment interview

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study sample includes students enrolled in the University of New Mexico (UNM), Department of Psychiatry and Behavioral Health Sciences CSC program. At the time of the study, the UNM CSC Program included separate clinics for patients diagnosed with clinical high risk for psychosis (CHRp) or FEP.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Crisanti, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norman R, Malla A. Course of Onset and Relapse Schedule: Interview and Coding Instruction Guide.; 2002. Prevention and Early Intervention for Psychosis Program. Available from author.
- [Background] Topkaya N, Sahin E, Meydan B. The Development, Validity, and Reliability of the Barriers to Seeking Psychological Help Scale for College Students. Int J High Educ. 2017;6(1):48-62.

RESULTS

PARTICIPANT FLOW:
Groups:
- Students Enrolled In Coordinated Specialty Care: The number of students determined eligible for Coordinated Specialty Care that were originally screened through the PQ-B at the college counseling center. This is a feasibility study so no intervention was administered.
Period: Overall Study
Arm/Group | Students Enrolled In Coordinated Specialty Care
Started | 25
Completed | 24
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Data are only available for 24 participants because after one participant was consented to participate in the study, they needed to reschedule and then did not show up for their interview
Groups:
- Students Enrolled in Coordinated Specialty Care: Students Enrolled In Coordinated Specialty Care that were originally identified through the PQ-B screen implemented in the college counseling center
Arm/Group | Students Enrolled in Coordinated Specialty Care
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.4 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Duration of Untreated Psychosis
Description: Duration of Untreated Psychosis determined upon enrollment to coordinated specialty care
Time Frame: Measured upon admission (baseline) to coordinated specialty care (CSC)
Population: 17 of the participants were determined to be at clinical high risk of psychosis rather than experiencing first episode psychosis. Duration of untreated psychosis can not be determined for participants at clinical high risk of psychosis. The other seven participants were determined to be experiencing their first episode of psychosis however were missing data on duration of psychosis.
Arm/Group | Students Enrolled in Coordinated Specialty Care
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Steps to Coordinated Specialty Care
Description: Measured among those who meet criteria for first episode psychosis or clinical high risk using the Circumstances of Onset and Relapse Schedule, and is operationalized as the number of steps between the onset of symptoms and admission to CSC for first episode psychosis or clinic high risk. The CORS includes the Topography of Psychotic Episode (TOPE), which traces the process of seeking treatment by identifying step-by-step contacts with medical, mental health, and/or community services in the pathway toward enrollment in CSC. Participants were asked if they had ever sought out a particular service or professional for mental health problems, and if so, the approximate date of that encounter.
Time Frame: Measured upon admission (baseline) to coordinated specialty care (CSC)
Measure: Mean (Standard Deviation); unit: Number of contacts prior to CSC
Groups:
- Participants Enrolled In Coordinated Specialty Care: The number of students determined eligible for Coordinated Specialty Care that were originally screened through the PQ-B at the college counseling center.
Arm/Group | Participants Enrolled In Coordinated Specialty Care
Number analyzed (Participants) | 24
Number of contacts prior to CSC | 5.71 (3.70)

3. Secondary Outcome: Perceived Barriers to Seeking Psychological Help
Description: Measured among those who meet criteria for first episode psychosis or clinical high risk by the Barriers to Seeking Psychological Help Scale (BSPHS), developed to measure barriers related to psychological help-seeking for college students. The self-report scale includes 17 items rated on a five point scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The scale includes five subscales: (1) fear of being stigmatized by society, (2) trust in the mental health professional, (3) difficulties in self-disclosure, (4) perceived devaluation, and, (5) lack of knowledge. BSPHS total score and scores for all subscales are determined by taking the mean of responses to all items for the entire scale and the mean of responses for each subscale, respectively. Higher scores indicate higher perceived barriers for the entire scale and all subscales.
Time Frame: Measured upon admission (baseline) to coordinated specialty care (CSC).
Population: Student enrolled in Coordinated Specialty Care that completed the Barriers to Seeking Psychological Help Scale
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Students Enrolled in Coordinated Specialty Care: Number of Students Enrolled in Coordinated Specialty Care that were identified via the PQ-B screen for early psychosis at the college counseling center
Arm/Group | Students Enrolled in Coordinated Specialty Care
Number analyzed (Participants) | 24
score on a scale
  Total Perceived Barriers to Care Mean Score | 2.58 (0.55)
  Fear of being stigmatized by society subscale mean score | 2.68 (0.85)
  Trust in the mental health professional subscale mean score | 2.70 (0.69)
  Difficulties in self-disclosure subscale mean score | 2.57 (0.91)
  Perceived devaluation subscale mean score | 2.39 (0.94)
  Lack of knowledge subscale mean score | 2.51 (0.83)

ADVERSE EVENTS:
Time Frame: This was not a follow-up study, data were only collected at baseline.
Groups:
- Number of Students Enrolled in Coordinated Specialty Care: Number of students enrolled in coordinated specialty care after being screened for early psychosis using the PQ-B at the college counseling center
Arm/Group | Number of Students Enrolled in Coordinated Specialty Care
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT03983421/Prot_SAP_000.pdf